CLINICAL TRIAL: NCT06142656
Title: Efficacy of Vildagliptin Versus Metformin in Poly Cystic Ovary Syndrome: A Randomized Clinical Trial
Brief Title: Efficacy of Vildagliptin Versus Metformin in Poly Cystic Ovary Syndrome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, engy wahsh, LECTURER OF CLINICAL PHARMACY, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRC-Ph-2307004
Record Dates: First submitted 2023-11-13; First posted 2023-11-21 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Poly Cystic Ovary Syndrome
MeSH Terms: interventions — Metformin; Vildagliptin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin Hydrochloride tablet
- Vildagliptin (Active Comparator)
  Interventions: Drug: Vildagliptin 50 MG

INTERVENTIONS:
Drug: Metformin Hydrochloride tablet — Metformin Hydrochloride 850 mg oral tablet
  Arms: Metformin
Drug: Vildagliptin 50 MG — Vildagliptin 50 MG oral tablets
  Arms: Vildagliptin

SUMMARY:
Polycystic ovary syndrome (PCOS) is an endocrine disorder that affects approximately 10-20% of women of reproductive age, Management strategies for PCOS include lifestyle modifications such as diet and physical activity that are the first-line approach to treatment; however, they are reported to be minimally effective in reducing weight or treating PCOS-related symptoms.Pharmacological options are also available; however, they are not explicitly approved for PCOS treatment as they have been primarily used to treat other conditions such as T2DM

ELIGIBILITY:
Inclusion Criteria:

-Women diagnosed with PCOS according to Rotterdam 2003 criteria National Institute of Health criteria.

Exclusion Criteria:

* Patients with history of diabetes mellitus (Type 1 or 2).
* Patients with liver or renal dysfunction; inflammatory diseases; autoimmune disease; cancer, acute cardiovascular event within last three months
* Known hypersensitivity or contraindications to use dipeptidyl peptidase-4 (DPP-4) inhibitors
* Eating disorders (anorexia, bulimia) or gastrointestinal disorders

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of luteinizing hormone (LH) | at baseline and after 3 months
  serum luteinizing hormone (LH)
Concentration of Follicle-stimulating hormone | at baseline and after 3 months
  Serum Follicle-stimulating hormone
Concentration of Free androgen index | at baseline and after 3 months
  serum Free androgen index
Concentration of total testosterone | at baseline and after 3 months
  serum total testosterone

CONTACTS AND LOCATIONS:
Overall Officials: ahmed hussein, PhD, Principal Investigator — october 6 university hospital
Locations (1):
- October 6 university hospital, Giza, Egypt